CLINICAL TRIAL: NCT04656275
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Different Oral Doses of BI 1323495 Bid Versus Placebo in Patients With Non-cystic Fibrosis Bronchiectasis (Randomised, Double-blind, Placebo-controlled, Parallel Group Trial)
Brief Title: A Study in Patients With Non-cystic Fibrosis Bronchiectasis to Test How Well Different Doses of BI 1323495 Are Tolerated and How BI 1323495 Affects Biomarkers of Inflammation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1405-0008; 2019-003853-27 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1323495 treatment group (part 1) (Experimental): Part 1
  Interventions: Drug: BI 1323495
- BI 1323495 treatment group (part 2) (Experimental): Part 2
  Interventions: Drug: BI 1323495
- Placebo group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1323495 — BI 1323495
  Arms: BI 1323495 treatment group (part 1); BI 1323495 treatment group (part 2)
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study is open to adults with non-cystic fibrosis bronchiectasis. The main purpose of this study is to find out how a medicine called BI 1323495 is tolerated by people with non-cystic bronchiectasis.

The study tests 2 different doses of BI 1323495. Some of the participants get placebo. It is decided by chance who gets BI 1323495 and who gets placebo. Participants take BI 1323495 or placebo as tablets twice a day for 3 months. Placebo tablets look like BI 1323495 tablets but do not contain any medicine. Participants can also continue taking standard medicines for noncystic bronchiectasis throughout the study.

Participants are in the study for about 4 months. During this time, the participants visit the study site about 11 times and get about 2 phone calls. At the visits, doctors check the health of the participants and note any health problems that could have been caused by BI 1323495.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 80 years (inclusive) at the time of informed consent signature, male and female (not of childbearing potential) subjects

  --For 'female not of childbearing potential' at least one of the following criteria must be fulfilled:
  * Permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy; tubal ligation is not a method of permanent sterilisation)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea without an alternative medical cause (in questionable cases a blood sample with Follicle Stimulating Hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory).
  * Men must be vasectomised with documented absence of sperm or use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after the last administration of trial medication if their sexual partner is a woman of childbearing potential (WOCBP)
* Clinical history consistent with non cystic fibrosis bronchiectasis (nCFB) (cough, chronic sputum production and/or recurrent respiratory infections) and proven and documented diagnosis of bronchiectasis by computed tomography (CT) scan including dilated airways compatible with bronchiectasis at initial diagnosis. Bronchiectasis of various etiologies will be allowed, with exclusion criteria as below.
* Vaccination against Streptococcus pneumoniae in accordance with national vaccination recommendations
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation.
* FEV1 ≥ 30 % predicted (post-bronchodilator) at Screening Visit 1.
* Stable (i.e., no dose change) regimen of standard nCFB treatment (including - but not limited to - hypertonic inhalation solutions, mucolytics, Long Acting Muscarinic Agonists (LAMA)/ Long Acting Beta Agonists (LABA) / inhaled corticosteriods (iCS), oral antibiotic maintenance regimen, and physiotherapy), if applicable, administered at least for 4 weeks prior to Screening Visit 1 and throughout the run-in period.
* Regular daily sputum producers with a history of chronic expectoration who are able to provide a typical bronchiectasis sputum sample at Screening Visit 1.
* Sputum neutrophil elastase positive based on point of care test (NEATstik® score ≥ 6) assessment at Visit 2a and Visit 2b.
* Subjects genotyped as UDP-Glucuronosyltransferase-2B17 (UGT2B17) extensive metabolizers prior to randomisation, i.e., carrying at least one functional allele of the UGT2B17 gene (*1/*1 or *1/*2)

Exclusion Criteria:

* Any finding in the medical examination (including BP, pulse rate (PR), or ECG) and/or laboratory value and/or any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Concomitant diagnosis of pulmonary disease other than bronchiectasis, chronic obstructive pulmonary disease (COPD), or asthma.
* A current diagnosis of cystic fibrosis (CF), primary immunodeficiency, active Allergic Bronchopulmonary Aspergillosis (ABPA) (defined by receipt of corticosteroids, anti-fungal treatment or monoclonal antibody treatment), or alpha-1 antitrypsin (A1AT) deficiency as underlying disease.
* A history or current immunodeficiency or are currently being treated (or are planned to be treated) with immunomodulatory drugs (except for iCS or low-dose oral corticosteroids), including disease-modifying anti-rheumatic drugs (DMARDs), and/or Immunglobulin G (IgG) treatments. Other medication that is excluded will be provided in the investigator site file (ISF). On the day of the site visit with lung function measurement, no bronchodilators should be used until after completion of lung function assessment
* Any acute infections defined as infections requiring antibiotic therapy, or Upper Respiratory Tract Infection (URTI). Are currently being treated (or are planned to be treated) for a nontuberculous mycobacterial (NTM) lung infection or tuberculosis.
* A history of invasive pneumococcal disease.
* Inhaled antibiotic treatment or cycling oral antibiotic treatment with changed dose regimen 4 weeks prior to Screening Visit 1.
* A treatment for a pulmonary exacerbation 4 weeks prior to Screening Visit 1.
* Laboratory confirmed severe acute respiratory syndrome (SARS)-coronavisurs (CoV)-2 infection (PCR positive) within 4 weeks prior to Screening Visit 1.
* Household contact with an individual with confirmed SARS-CoV-2 infection within 4 weeks prior to Screening Visit 1.
* Further exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double blind, placebo-controlled, parallel group design, to compare safety and tolerability of different doses of BI 1323495 with placebo and to assess pharmacodynamics of BI 1323495 in sputum and in blood as well as early signs of clinical efficacy of BI 1323495 in patients with non-cystic fibrosis bronchiectasis (nCFB).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Part A: Placebo Bid: This arm comprises all placebo treated participants in trial part A. Participants were randomized in the dose group in a 3:1 ratio (test treatment to placebo). Participants were administered for 12 weeks, twice a day (bid) an oral dose of film-coated tablets of matching placebo (the matching placebo was mannitol, microcrystalline cellulose, and magnesium stearate) together with about 240 milliliter (mL) of water. The doses were taken after 15-30 minutes (min) of food intake including a fat component. Evening and morning dose were taken with a 12 hours (h) time interval approximately at the same time each day during the treatment phase, within a time window of +/- 1 hour.
- Part A: 30 mg BI 1323495 Bid: 3 film-coated tablets of 10 milligram (mg) BI 1323495 were administered orally twice daily (bid) (total dose: 60 mg) together with about 240 milliliter of water over 12 weeks. The doses were taken after 15-30 min of food intake including a fat component. Evening and morning dose were taken with a 12 h time interval approximately at the same time each day during the treatment phase, within a time window of +/- 1 hour.
Period: Overall Study
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Started | 2 | 5
Completed (Completed treatment) | 0 | 1
Not Completed | 2 | 4
Not completed — Study terminated by sponsor | 2 | 4

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (8.5) | 59.2 (5.3) | 57.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Absolute neutrophil elastase (NE) activity in sputum [Mean (Standard Deviation); unit: Relative fluorescence unit (RFU)] — The Absolute neutrophil elastase (NE) activity in sputum baseline values were calculated as the mean of the baseline values (at day -6, -2, day 1 predose). Relative fluorescence unit (RFU) is the standard output of a florescence reader. RFU (ex 360 nm, em460 nm). Population: Only patients with no missing values for absolute neutrophil elastase (NE) activity in sputum are reported.
  Relative fluorescence unit (RFU)
    number analyzed (Participants) | 2 | 4 | 6
    (all) | 19115.0 (598.2) | 15610.4 (9991.7) | 16778.6 (7952.8)
Neutrophil cell count in sputum [Mean (Standard Deviation); unit: Neutrophils*10^9/Liter] — Neutrophil cell count in sputum baseline values were calculated as the mean of the baseline values (at day -6, -2, day 1 predose). RUF: Relative fluorescence unit Population: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments.
  Neutrophils*10^9/Liter
    number analyzed (Participants) | 2 | 4 | 6
    (all) | 338.9 (40.7) | 322.0 (123.9) | 327.6 (98.0)
NE activity in whole blood after stimulation with zymosan, normalized to neutrophil counts [Mean (Standard Deviation); unit: RFU/(10^9 cells/L)] — NE activity in whole blood after stimulation with zymosan, baseline values were measured at Day 1, 2.5 hours (hrs) prior first treatment administration.
  Relative fluorescence unit (RFU) is the standard output of a florescence reader. RFU (ex 360 nm, em460 nm).
  RFU/(10^9 cells/L) | 5354.8 (3506.7) | 7278.5 (2574.4) | 6728.9 (2710.9)
Absolute post-bronchodilator forced expiratory volume in one second, FEV1 [Mean (Standard Deviation); unit: Milliliter (mL)] — Absolute post-bronchodilator forced expiratory volume in one second (FEV1) baseline values were measured at Day -2.
  Milliliter (mL) | 3052.5 (475.9) | 2177.2 (434.5) | 2427.3 (588.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: Number of participants with drug-related adverse events (AEs) is presented. Participants with treatment-emergent drug-related Adverse Events (AEs) is reported.
Time Frame: From drug administration until 12:00 AM on day after last administration of study drug + 7 days residual effect period (REP) or 12:00 AM on day after last contact date, which ever occurs first. Up to 13 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Number analyzed (Participants) | 2 | 5
Participants | 0 | 2

2. Secondary Outcome: Change From Baseline to Day 15, Day 29, Day 57, Day 78, Day 82 and Day 98 in Absolute Neutrophil Elastase (NE) Activity in Sputum
Description: The change from baseline to Day 15, Day 29, Day 57, Day 78, Day 82 and Day 98 in absolute neutrophil elastase (NE) activity in sputum is reported. The baseline value was calculated as the mean of the baseline values (at day -6, -2, day 1 predose). RFU is the standard output of a florescence reader. RFU (ex 360 nm, em460 nm).
Time Frame: At baseline Day -6, Day -2, Day 1 before the first dose and at Day 15, Day 29, Day 57, Day 78, Day 82 and Day 98.
Population: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments. Only patients with no missing values for absolute neutrophil elastase (NE) activity in sputum are reported.
Measure: Mean (Standard Deviation); unit: Relative fluorescence unit (RFU)
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Number analyzed (Participants) | 2 | 5
Relative fluorescence unit (RFU)
  Change from baseline to Day 15: number analyzed (Participants) | 1 | 3
  Change from baseline to Day 15 | 3301.0 | -156.9 (2028.5)
  Change from baseline to Day 29: number analyzed (Participants) | 1 | 3
  Change from baseline to Day 29 | 2745.0 | -194.4 (660.6)
  Change from baseline to Day 57: number analyzed (Participants) | 0 | 3
  Change from baseline to Day 57 |  | -497.1 (217.9)
  Change from baseline to Day 78: number analyzed (Participants) | 1 | 0
  Change from baseline to Day 78 | 1665.0 |
  Change from baseline to Day 82: number analyzed (Participants) | 0 | 1
  Change from baseline to Day 82 |  | 383.0
  Change from baseline to Day 98: number analyzed (Participants) | 0 | 2
  Change from baseline to Day 98 |  | 582.3 (1257.7)

3. Secondary Outcome: Change From Baseline to Week 12 (at Week 2, Week 4, Week 8, Week 12) in Neutrophil Cell Count in Sputum
Description: The change from baseline to week 12 (at Week 2, Week 4, Week 8, Week 12) in absolute neutrophil cell count in sputum is reported. The baseline value was calculated as the mean of the baseline values (at day -6, -2, day 1 predose).
  RFU: Relative fluorescence unit
Time Frame: At baseline Day -6, Day -2, Day 1 before the first dose and at at Week 2, Week 4, Week 8, Week 12 during treatment.
Population: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments. Only patients with no missing values for neutrophil cell count in sputum are reported.
Measure: Mean (Standard Deviation); unit: Neutrophils*10^9/Liter
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Number analyzed (Participants) | 2 | 4
Neutrophils*10^9/Liter
  Time-matched change from baseline to Week 2: number analyzed (Participants) | 1 | 4
  Time-matched change from baseline to Week 2 | -9.7 | 27.1 (82.9)
  Time-matched change from baseline to Week 4: number analyzed (Participants) | 1 | 3
  Time-matched change from baseline to Week 4 | 16.8 | -7.8 (11.3)
  Time-matched change from baseline to Week 8: number analyzed (Participants) | 0 | 3
  Time-matched change from baseline to Week 8 |  | 9.7 (23.4)
  Time-matched change from baseline to Week 12: number analyzed (Participants) | 1 | 1
  Time-matched change from baseline to Week 12 | -47.7 | 69.5

4. Secondary Outcome: Change From Baseline to Week 12 in Neutrophil Elastase (NE) Activity in Whole Blood After Stimulation With Zymosan (Normalized to Neutrophil Counts)
Description: The change of NE activity from baseline to Day 15, Day 29, Day 57, Day 78, Day 82 and Day 98 in whole blood after stimulation with zymosan (normalized to neutrophil counts) is reported.
  Relative fluorescence unit (RFU) is the standard output of a florescence reader. RFU (ex 360 nm, em460 nm).
Time Frame: At baseline Day 1, 2.5 hours (hrs) before the first dose and at Day 15, Day 29, Day 57, Day 78, Day 82 and Day 98.
Population: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments. Only patients with no missing values for Neutrophil Elastase (NE) activity in whole blood after stimulation with zymosan are reported.
Measure: Mean (Standard Deviation); unit: RFU/(10^9 cells/L)
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Number analyzed (Participants) | 2 | 5
RFU/(10^9 cells/L)
  Time-matched change from baseline to Day 15: number analyzed (Participants) | 1 | 4
  Time-matched change from baseline to Day 15 | 95.8 | -7733.9 (2153.2)
  Time-matched change from baseline to Day 29 / -2:30: number analyzed (Participants) | 1 | 3
  Time-matched change from baseline to Day 29 / -2:30 | 99.2 | -6306.0 (852.6)
  Time-matched change from baseline to Day 29 / 6:00: number analyzed (Participants) | 1 | 3
  Time-matched change from baseline to Day 29 / 6:00 | 238.1 | -6649.6 (1505.1)
  Time-matched change from baseline to Day 57: number analyzed (Participants) | 1 | 2
  Time-matched change from baseline to Day 57 | -630.3 | -5889.9 (786.0)
  Time-matched change from baseline to Day 82: number analyzed (Participants) | 2 | 3
  Time-matched change from baseline to Day 82 | -622.6 (1089.0) | -5689.9 (3610.3)
  Time-matched change from baseline to Day 98 | -326.4 (1295.0) | 1221.1 (2703.8)

5. Secondary Outcome: Change From Baseline to Week 12 in Absolute Post-bronchodilator Forced Expiratory Volume in One Second, FEV1
Description: The change from baseline to week 12 (at Week 2, Week 8, Week 12) in absolute post-bronchodilator forced expiratory volume in one second (FEV1).
Time Frame: At baseline Day -2 before the first dose and at at Week 2, Week 8, Week 12 during treatment.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
Number analyzed (Participants) | 2 | 5
Milliliter (mL)
  Time-matched change from baseline to Week 2 | 38 (113.1) | 1.4 (78.6)
  Time-matched change from baseline to Week 8: number analyzed (Participants) | 1 | 3
  Time-matched change from baseline to Week 8 | -27.0 | 1.0 (220.1)
  Time-matched change from baseline to Week 12: number analyzed (Participants) | 1 | 2
  Time-matched change from baseline to Week 12 | -138.0 | -40.0 (178.2)

ADVERSE EVENTS:
Time Frame: From drug administration until 12:00 AM on day after last administration of study drug + 7 days (REP) or 12:00 AM on day after last contact date, which ever occurs first. Up to 13 weeks. All-cause mortality: Up to 13 weeks.
Description: Treated set (TS): The treated set included all patients who were randomised and received at least one dose of study drug. The treatment assignment was determined based on the first actual treatment the patients received. The TS was used for safety analyses and evaluation of biomarker and clinical assessments.
Arm/Group | Part A: Placebo Bid | Part A: 30 mg BI 1323495 Bid
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo Bid (N=2) | Part A: 30 mg BI 1323495 Bid (N=5)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Part B of the study was not started due to the same reason that caused discontinuation of Part A, i.e. due to the need to clarify findings in nonclinical toxicity testing in animals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04656275/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04656275/SAP_001.pdf